CLINICAL TRIAL: NCT00714337
Title: A Phase I, Single-Centre, Randomised, Open-Label, Five-Way Cross-Over Formulation- and Food-Effect Study in Healthy Volunteers to Assess the Pharmacokinetics of AZD1386 After Single Doses of Two Oral Solid Formulations and an Oral Solution
Brief Title: Formulation and Food Effect Study of AZD1386 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD PhD. Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5090C00007; EudraCT 2008-002150-37
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Pharmacokinetics
Keywords: Formulation; pharmacokinetics
MeSH Terms: interventions — AZD1386

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): fasting state
  Interventions: Drug: AZD1386
- 2 (Experimental): fasting state
  Interventions: Drug: AZD1386
- 3 (Experimental): non-fasting state
  Interventions: Drug: AZD1386
- 4 (Experimental): fasting state
  Interventions: Drug: AZD1386
- 5 (Experimental): non-fasting state
  Interventions: Drug: AZD1386

INTERVENTIONS:
Drug: AZD1386 — One single oral dose of 90mg (36mL of AZD1386 2.5mg/mL oral solution).
  Arms: 1
Drug: AZD1386 — One single oral dose of 90mg (3 x 30mg AZD1386 capsules)
  Arms: 2; 3
Drug: AZD1386 — One single oral dose of 90mg (6 x 15mg AZD1386 tablets)
  Arms: 4; 5

SUMMARY:
To investigate the pharmacokinetics of two oral solid formulations of AZD1386 in relation to the AZD1386 oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-fertile (Amenorrhea and no pregnancy in the last 12 months prior to enrolment or documentation of being irreversible surgically sterile).
* Healthy male volunteers with BMI between 18 and 30 kg/m2
* Clinical normal physical findings, including blood pressure, pulse rate above 45 bpm, ECG, and laboratory assessments.
* Normal QTc interval on baseline ECG, between 360-450 msec, according to the Fridericia formula.

Exclusion Criteria:

* History of severe allergy/hypersensitivity or symptoms/signs of ongoing allergy/hypersensitivity as judged by the Investigator.
* Requirement of concomitant medication during the study, excluding hormone replacement therapy (HRT) or use of drugs with enzyme inducing properties with 3 weeks of first dose
* Smoking more than 7 cigarettes per week or consumption of more than 3 portion of snuff or equivalent per day within 30 days before first administration of study drug
* A family history of short QT syndrome (SQTS) or sudden cardiac death (SCD) amongst first degree relatives and who have a QT/QTc <360 ms

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during study days

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Francke, MD, Principal Investigator — PAREXEL Clinical Pharmacology Research Unit